CLINICAL TRIAL: NCT02241408
Title: Autologous Adipose Stromal Vascular Fraction Outcomes in Osteoarthritis Research Study
Brief Title: Outcomes Data of Adipose Stem Cells to Treat Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: StemGenex (Industry)
Responsible Party: Sponsor
Other Study IDs: SVF01OA; ASCOA-01
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the impact that treatment with a cellular concentrate derived from an individual's own fat, known as the stromal vascular fraction (SVF), has on joint pain and functionality in people with Osteoarthritis (OA). SVF contains components with "regenerative" properties, including stem cells that have shown promise for ameliorating specific disease conditions. This study is designed to evaluate joint pain and functionality changes in individuals with OA for up to 12 months following SVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Over the age of 18
* Diagnosed with OA of the knee and/or hip
* Scheduled for intravenous and intra-articular administrations of autologous SVF
* Capable of understanding and willing to sign informed consent
* Willing and able to complete brief phone interviews
* Willing and able to complete online surveys

Exclusion Criteria:

* Co-morbidity with an autoimmune disorder
* Pregnant, may become pregnant, or breastfeeding
* Subjects for which baseline data is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Knee Assessment Over the Course of a 12 Month Period as Measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) | Baseline, 12 months
  The change from baseline over the course of 12 months using participants' assessment of their knee and associated problems. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 3, 6, and 12). Answer options are graded on a 5 point Likert scale and each question gets a score from 0 to 4.
Change from Baseline in Overall Hip Assessment Over the Course of a 12 Month Period as Measured by the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) | Baseline, 12 months
  The change from baseline over the course of 12 months using participants' assessment of their hip and associated problems. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 3, 6, and 12). Answer options are graded on a 5 point Likert scale and each question gets a score from 0 to 4.

SECONDARY OUTCOMES:
Change from Baseline in Knee Pain at Month 12 as Measured by Participants Using the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) The Pain Subscale | Baseline, Month 12
  Participant assessment in the change in knee pain from baseline to month 12 using the KOOS pain subscale.
Change from Baseline in Function in Daily Living (ADL) at Month 12 as Measured by Participants Using the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) The ADL Subscale | Baseline, Month 12
  Participant assessment in the change in function in daily living from baseline to month 12 using the KOOS ADL subscale.
Change from Baseline in Function in Sport and Recreation at Month 12 as Measured by Participants Using the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) The Sport/Rec Subscale | Baseline, Month 12
  Participant assessment in the change in sport and recreation from baseline to month 12 using the KOOS sport/rec subscale.
Change from Baseline in Knee Related Quality of Life (QOL) at Month 12 as Measured by Participants Using the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) The Knee Related Quality of Life Subscale | Baseline, Month 12
  Participant assessment in the change in knee related quality of life from baseline to month 12 using the KOOS QOL subscale.
Change from Baseline in Other Knee Symptoms at Month 12 as Measured by Participants Using the Knee Injury and Osteoarthritis Outcome Score (KOOS LK 1.0) The Other Symptoms Subscale | Baseline, Month 12
  Participant assessment in the change in other knee symptoms from baseline to month 12 using the KOOS other symptoms subscale.
Change from Baseline in Hip Pain at Month 12 as Measured by Participants Using the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) The Pain Subscale | Baseline, Month 12
  Participant assessment in the change in hip pain from baseline to month 12 using the HOOS pain subscale.
Change from Baseline in Function in Daily Living (ADL) at Month 12 as Measured by Participants Using the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) The ADL Subscale | Baseline, Month 12
  Participant assessment in the change in function in daily living from baseline to month 12 using the HOOS ADL subscale.
Change from Baseline in Function in Sport and Recreation at Month 12 as Measured by Participants Using the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) The Sport/Rec Subscale | Baseline, Month 12
  Participant assessment in the change in function in sport and recreation from baseline to month 12 using the HOOS sport/rec subscale.
Change from Baseline in Hip Related Quality of Life (QOL) at Month 12 as Measured by Participants Using the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) The QOL Subscale | Baseline, Month 12
  Participant assessment in the change in hip related quality of life from baseline to month 12 using the HOOS QOL subscale.
Change from Baseline in Other Hip Symptoms at Month 12 as Measured by Participants Using the Hip Dysfunction and Osteoarthritis Outcome Score (HOOS LK 2.0) The Other Symptoms Subscale | Baseline, Month 12
  Participant assessment in the change in other hip symptoms from baseline to month 12 using the HOOS other symptoms subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- StemGenex, San Diego, California, United States